CLINICAL TRIAL: NCT02667600
Title: Study Assessing Blood Loss Measurement During Cesarean Delivery With Triton Device
Brief Title: Blood Loss Measurement During Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Alex James Butwick (Other)
Responsible Party: Sponsor-Investigator, Alex James Butwick, Assistant Professor of Anesthesiology, Perioperative and Pain Medicine (OB), Stanford University
Organization: Stanford University (Other)
Other Study IDs: 35648
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Pregnancy
Keywords: Cesarean; Blood Loss; Triton
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cesarean Section Group: Patients undergoing cesarean section

SUMMARY:
The aim of this study is to assess the ability of the Triton Device to measure blood loss among women undergoing elective and non-elective cesarean delivery. This patient population often experiences significant blood loss during surgery, and measurements of surgical blood loss are often inaccurate.

DETAILED DESCRIPTION:
This is an observational study. Potential participants will be approached by a member of the research team prior to surgery. Healthy ASA 1, 2, or 3 patients undergoing uncomplicated Cesarean delivery will be recruited. The Triton device will be used during the surgery to estimate blood loss. Specifically, the device takes pictures of the blood saturated laps and fluid collection canister and calculates hemoglobin loss and overall blood loss.

Serum hemoglobin samples will be collected at baseline on presentation to the pre-operative area, within 15 mins of arrival in PACU and at 24 hrs post cesarean delivery. Blood sampling will take place by venipuncture technique from a vein in the arm. Maternal vital signs during the perioperative period (heart rate, maternal mean arterial blood pressure, anesthetic technique, fluid administration, and surgical data will be recorded.

All patient will have a neuraxial anesthetic of a spinal or combined spinal/epidural. Fluid administration will be under the discretion of the anesthesiologist and will follow standard guidelines including 1L of Lactated Ringers co-load at time of spinal and 1-2L of crystaloid intraoperatively.

At the end of the cesarean section, the following measurements will be made:

1. tEBL: Triton device will be used to measure blood loss on wet and dry soaked laps and in the suction canister. These measurements will be used to calculate tEBL.
2. vEBL: The attending obstetrician and anesthesiologist will independently be asked to provide estimates for total blood loss (vEBL). We will use both values in separate regression analyses
3. qEBL: Blood loss will be measured by cumulative measurement of the following: the volume of blood in the suction chamber at the end of surgery (and subtracting the estimated amniotic fluid from the suction chamber; weight of blood soaked laps; estimated spillage of blood (in ml) in and around the surgical field (not collected on laps or in suction chamber).

Using mixed effects modeling, we will determine whether estimated blood loss measurements using Triton (tEBL) can be used to predict postpartum hemoglobin (Hb) levels, after accounting for the predelivery Hb level, intraoperative intravenous fluids and patient/operative factors.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class I-III
* undergoing Cesarean delivery under neuraxial anesthesia
* age between 18 and 50
* gestational age greater than or equal to 37 completed weeks
* all ethnicities

Exclusion Criteria:

* contraindication for epidural or spinal analgesia (bleeding diathesis, neuropathy, severe scoliosis, local anesthetic allergy)
* inability to adequately understand the consent form

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy female patients undergoing uncomplicated Cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Difference in blood loss measurements | Day Of Surgery
  Compare blood loss estimates between the triton device, visual estimation of blood loss, and cumulative measurements of blood loss during a cesarean delivery

SECONDARY OUTCOMES:
Triton Blood Loss Prediction of Post Partum Hemoglobin | 24-48 hours post surgery
  Using mixed effects modeling, it will be determine whether estimated blood loss measurements using Triton (tEBL) can be used to predict postpartum hemoglobin (Hb) levels, after accounting for the predelivery Hb level, intraoperative intravenous fluids and patient/operative factors.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Butwick, FRCA, Principal Investigator — Stanford University; Brendan Carvalho, MBBCh, FRCA, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al Kadri HM, Al Anazi BK, Tamim HM. Visual estimation versus gravimetric measurement of postpartum blood loss: a prospective cohort study. Arch Gynecol Obstet. 2011 Jun;283(6):1207-13. doi: 10.1007/s00404-010-1522-1. Epub 2010 May 28. PMID 20508942
- [Background] Konig G, Holmes AA, Garcia R, Mendoza JM, Javidroozi M, Satish S, Waters JH. In vitro evaluation of a novel system for monitoring surgical hemoglobin loss. Anesth Analg. 2014 Sep;119(3):595-600. doi: 10.1213/ANE.0000000000000198. PMID 24806138
- [Background] Holmes AA, Konig G, Ting V, Philip B, Puzio T, Satish S, Waters JH. Clinical evaluation of a novel system for monitoring surgical hemoglobin loss. Anesth Analg. 2014 Sep;119(3):588-594. doi: 10.1213/ANE.0000000000000181. PMID 24797122
- [Derived] Fedoruk K, Seligman KM, Carvalho B, Butwick AJ. Assessing the Association Between Blood Loss and Postoperative Hemoglobin After Cesarean Delivery: A Prospective Study of 4 Blood Loss Measurement Modalities. Anesth Analg. 2019 May;128(5):926-932. doi: 10.1213/ANE.0000000000003449. PMID 29847380